CLINICAL TRIAL: NCT06357715
Title: Effectiveness of Neurodynamic Sliding Mobilisation in the "Slump" Position in Relation to the Perceptible Pain Threshold in Asymptomatic People, a Cross-over Randomised Controlled Trial
Brief Title: Effectiveness of Neurodynamic Sliding Mobilisation in the "Slump" Position in Relation to the Perceptible Pain Threshold in Asymptomatic People
Acronym: SPEAKER 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/0373/HP
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-01

CONDITIONS: Voluntary

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the second physiotherapist who evaluate the pressure pain
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neurodynamic sliding mobilisation in the "Slump" position (Active Comparator): "slump"position
  Interventions: Other: "slump"position; Other: no" slump" position
- mobilisation, out of the "Slump" position (Placebo Comparator): no "slump"position
  Interventions: Other: "slump"position; Other: no" slump" position

INTERVENTIONS:
Other: "slump"position — neurodynamic sliding mobilisation in the "slump" position
Other: no" slump" position — placebo

SUMMARY:
According to the French National Health Agency, the use of manual therapy techniques is "possible" [grade B] as part of a multimodal combination of treatments for low back pain. These include so-called "neurodynamic" neural mobilisations, which aim in particular to desensitise the pain system and activate descending inhibitory pathways, with effects on pain and function in patients with nerve-related low back pain. Most of the available evidence does not explain the mechanisms involved in neural mobilisation in the slump position. Pain reduction is observed in more areas of the body with sliding techniques than with traction techniques.

In this cross-over, randomised controlled trial, we therefore hypothesise that the neurodynamic sliding technique in the slump position acts on mechanisms linked to central pain modulation processes

ELIGIBILITY:
Inclusion Criteria:

Subjects aged 30 years or older and less than 65 years;

* Subjects considered naive to neurodynamic mobilisation techniques;
* Volunteers who have read and understood the information letter and have given their written consent to participate in the study;
* Fluent in spoken and read French;
* Effective contraception in women of childbearing age (progestin-only or intrauterine device or tubal ligation) for at least 12 months;
* For postmenopausal women, a confirmatory diagnosis must be obtained (non-drug-induced amenorrhoea for at least 12 months prior to the enrolment visit);
* Subject affiliated to a social security scheme.

Exclusion Criteria:

* Positive slump test on the day of the selection visit (production of asymmetric lumbar symptoms or painful radiations in at least one lower limb or unilateral reduction in physiological knee extension range of motion compared with the contralateral side);
* Neurological and neuropathic pain assessment score (DN4) greater than 4;
* Increase or decrease in sensory function in the lower limb compared with the contralateral side, as measured by Clinical Sensory Testing (CST);
* Any physical exertion of perceived intensity greater than 17 on the Borg 6-20 scale in the 72 hours prior to the trial and during the trial;
* Injury, complaint or symptom affecting the spine (cervical, thoracic, lumbar) and/or lower limb(s) requiring absence from work, school or leisure activities in the 12 months prior to enrolment;
* History of major surgery, injury to the trunk, spine and/or lower limb(s), or history of progressive rheumatic, neurological or oncological pathology;

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-11-06 (Estimated); Study Completion 2026-11-06 (Estimated)

PRIMARY OUTCOMES:
Difference in pressure at the moment when the volunteer indicates that the sensation of pressure becomes pain | immediately after the mobilisation and 1 day after the mobilisation
  Difference in pressure exerted on the territory of the sciatic nerve (gluteal region) at the moment when the volunteer indicates that the sensation of pressure becomes pain, on the dominant lower limb, between the same volunteer during two treatment sessions which differ only in the exposure to neurodynamic sliding mobilisation in the "Slump" position or to mobilisation outside the "Slump" position.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'investigation clinique CIC ROUEN, Rouen, France

IPD SHARING:
Plan to Share IPD: No